CLINICAL TRIAL: NCT04199403
Title: Assessment of Complication Risk Factors in a French National Cohort of Asplenic Patients
Acronym: SPLEEN
Status: Recruiting | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Collaborators: Pr Pierre BUFFET Institut National de la Transfusion Sanguine (Unknown); Dr Edouard TUAILLON Département Bactériologie-Virologie/INSERM U1058 CHU de Montpellier (Unknown)
Responsible Party: Sponsor
Other Study IDs: SPLEEN
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Asplenia
Keywords: spleen; asplenic patients; splenectomy; asplenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group

SUMMARY:
Spleen could have been surgically removed for trauma, cancer, auto-immune disease, or to perform a diagnosis. Spleen could be non-functional due to radiotherapy or splenic artery embolism. These patients are at risks of infectious diseases due to encapsulated bacteria, cancer, and thromboembolism disease. The purpose of this study is to assess complications occurring in French patients without spleen and to implement new diagnostic tools for follow-up.

DETAILED DESCRIPTION:
Asplenia can be congenital or acquired. Acquired asplenia can be due to diagnostic or therapeutic surgery, splenic artery embolization, or radiotherapy. Incidence of splenectomized patients was estimated between 10 and 15/100 000 persons in 2003. More recent data suggested a decrease in splenectomy due to increase of splenic artery embolization. From 212 to 2016, about 4000 splenectomy had still been performed.

Three different risks are known for asplenic patients: infectious, neoplastic, and thromboembolic. Prevalence rate of infectious complications in splenectomized patients was 3.2% with a mortality rate of 1.4%. A US cohort study including 8149 splenectomized veterans have shown that the risk of cancer was increased, so did the risk of thromboembolic disease, on a 27-year period of follow-up. Pathophysiology of these risks are not well known.

There are very few tools to assess splenic function: Howell-Jolly bodies in red blood cells, scintigraphy. These tools lack sensitivity and are not correlated with complications in asplenic patients.

To better understand how splenic function and how immunity evolves during time in asplenic patients, a longitudinal follow-up could be useful. There may be some differences between splenectomized patients, those who benefited from splenic artery embolization, and those who received radiotherapy. Infectious risk may be different between these three groups. Implementing new tools assessing residual splenic function could improve management of these patients. A prospective follow-up aims at accurately estimate the incidence rate of infectious and non-infectious complications in this population.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 year-old
* With asplenia due to splenectomy, splenic artery embolization or radiotherapy

Exclusion Criteria:

* Genetic asplenia including sick cell disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years with acquired asplenia due to splenectomy, artery embolization, or spleen radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of complication risk factors | 3 years
  Comparison between splenectomy and other type of asplenia for prevalence of infectious diseases, cancer, and thromboembolism disease

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu PUYADE, MD, Principal Investigator — C.H.U. de Poitiers
Locations (12):
- France (12):
  - C.H. d'Angoulême, Angoulême
  - C.H. Victor Dupouy, Argenteuil
  - C.H. de Béthune, Béthune
  - Hôpitaux de Chartres, Chartres
  - C.H.U. de Lille, Lille
  - C.H.U. de Montpellier, Montpellier
  - Hôtel-Dieu - CHU de Nantes, Nantes
  - C.H.U. de Poitiers, Poitiers
  - C.H.U. de Rouen, Rouen
  - C.H.U. de Toulouse, Toulouse
  - C.H. de Tourcoing, Tourcoing
  - C.H. de Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kristinsson SY, Gridley G, Hoover RN, Check D, Landgren O. Long-term risks after splenectomy among 8,149 cancer-free American veterans: a cohort study with up to 27 years follow-up. Haematologica. 2014 Feb;99(2):392-8. doi: 10.3324/haematol.2013.092460. Epub 2013 Sep 20. PMID 24056815
- [Result] Mebius RE, Kraal G. Structure and function of the spleen. Nat Rev Immunol. 2005 Aug;5(8):606-16. doi: 10.1038/nri1669. PMID 16056254
- [Result] Aiolfi A, Inaba K, Strumwasser A, Matsushima K, Grabo D, Benjamin E, Lam L, Demetriades D. Splenic artery embolization versus splenectomy: Analysis for early in-hospital infectious complications and outcomes. J Trauma Acute Care Surg. 2017 Sep;83(3):356-360. doi: 10.1097/TA.0000000000001550. PMID 28459796